CLINICAL TRIAL: NCT07388719
Title: A Prospective Interventional Study Comparing Standard and Dynamic Compliance-Guided Individualized Positive End-Expiratory Pressure on Intraoperative Oxygenation and Postoperative Pulmonary Complications in Obese Patients Undergoing Spinal Surgery
Brief Title: Comparison of Standard Versus Dynamic Compliance-Guided Individualized PEEP in Obese Patients Undergoing Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-2024-5206
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Postoperative Pulmonary Complications; Mechanical Ventilation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two parallel groups receiving either standard fixed PEEP or dynamic compliance-guided individualized PEEP during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard PEEP (Active Comparator): Patients assigned to this arm receive a fixed positive end-expiratory pressure (PEEP) of 5 cmH₂O throughout the intraoperative period during mechanical ventilation.
  Interventions: Device: Standard PEEP
- Dynamic Compliance-Guided Individualized PEEP (Experimental): Patients assigned to this arm receive individualized positive end-expiratory pressure (PEEP) titrated according to intraoperative dynamic lung compliance, with the aim of optimizing respiratory mechanics while avoiding overdistension.
  Interventions: Device: Standard PEEP

INTERVENTIONS:
Device: Standard PEEP — Application of a fixed positive end-expiratory pressure of 5 cmH₂O during intraoperative mechanical ventilation.

SUMMARY:
This study aims to compare standard positive end-expiratory pressure (PEEP) with dynamic compliance-guided individualized PEEP in obese patients undergoing elective spinal surgery under general anesthesia. Obesity and prone positioning during spinal surgery are associated with reduced lung compliance, atelectasis, and an increased risk of postoperative pulmonary complications.

Participants will be allocated to receive either a fixed standard PEEP or an individualized PEEP level determined according to intraoperative dynamic lung compliance. Intraoperative oxygenation, respiratory mechanics, arterial blood gas parameters, and hemodynamic variables will be assessed at predefined time points. Postoperative pulmonary complications within the first 24 hours after surgery will also be evaluated.

The study seeks to determine whether individualized PEEP titration based on dynamic compliance offers physiological or clinical advantages compared with a standard PEEP strategy in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years
* Body mass index (BMI) ≥30 kg/m²
* Scheduled for elective spinal surgery under general anesthesia
* Requirement for intraoperative mechanical ventilation
* American Society of Anesthesiologists (ASA) physical status II-III
* Provision of written informed consent

Exclusion Criteria:

* Pre-existing severe pulmonary disease (e.g., COPD GOLD stage III-IV, restrictive lung disease)
* Severe cardiac disease (e.g., heart failure with reduced ejection fraction, significant valvular disease)
* History of thoracic surgery affecting lung mechanics
* Pregnancy
* Emergency surgery
* Intraoperative need for deviation from the planned ventilation protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Intraoperative Oxygenation (PaO₂/FiO₂ Ratio) | From induction of anesthesia until the end of surgery
  The primary outcome is intraoperative oxygenation assessed by the arterial partial pressure of oxygen to fraction of inspired oxygen (PaO₂/FiO₂) ratio during mechanical ventilation.

SECONDARY OUTCOMES:
Dynamic Lung Compliance | From induction of anesthesia until the end of surgery
  Dynamic lung compliance (mL/cmH₂O) measured intraoperatively via ventilator respiratory mechanics monitoring.
Static Lung Compliance | From induction of anesthesia until the end of surgery
  Static lung compliance (mL/cmH₂O) measured intraoperatively via ventilator plateau pressure analysis.
Peak Airway Pressure | From induction of anesthesia until the end of surgery
  Peak inspiratory airway pressure (cmH₂O) measured intraoperatively using ventilator monitoring.
Plateau Airway Pressure | From induction of anesthesia until the end of surgery
  Plateau airway pressure (cmH₂O) measured intraoperatively during mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No